# **COVER PAGE**

Official Title: Mn/QD-SAC-Guided NIR-IIb Imaging and Antioxidant Therapy for

Ischemia-Reperfusion Injury in DIEP Flaps

Document Type: Study Protocol and Statistical Analysis Plan

ClinicalTrials.gov Identifier (NCT Number): NCTXXXXXXXX

Sponsor/Institution: Hubei Cancer Hospital

Study Location: Breast Surgery Department, Hubei Cancer Hospital, Wuhan, China

Principal Investigator: Xinhong Wu, MD

Department: Breast Surgery

Document Date: 11 Sep 2025

Version: v1.0

#### 1. SYNOPSIS

- (1) Background: Deep inferior epigastric perforator (DIEP) flap breast reconstruction is valuable but prone to microcirculatory instability and ischemia–reperfusion injury (I/R). NIR-IIb (1500–1700 nm) imaging offers deeper penetration and higher SNR than conventional ICG-NIR, potentially enabling earlier detection of perfusion deficits. A manganese-modified single-atom catalyst on NIR-IIb quantum dots (Mn/QD-SAC) combines deep-tissue imaging with broad-spectrum ROS-scavenging enzyme-mimetic activity to mitigate I/R damage.
- (2) Hypothesis: Intraoperative and postoperative application of Mn/QD-SAC will enable earlier and deeper detection of perfusion deficits via NIR-IIb imaging and attenuate ROS-driven inflammatory cascades, reducing adipose necrosis and partial flap loss.
- (3) Design: Preclinical materials development; in vitro mechanistic assays; small-animal DIEP-like flap I/R model for imaging/therapy; and an observational, minimal-risk human biospecimen sub-study (peripheral blood from DIEP patients) to assess circulating biomarkers.
- (4) Primary Endpoints: Flap survival rate at postoperative Day 7; NIR-IIb SNR and correlation with final flap survival area.
- (5) Secondary Endpoints: Materials properties; in vitro cell survival/apoptosis/ROS and cytokines; in vivo oxidative stress, inflammation, apoptosis, histology; safety and biodistribution.
- (6) Statistics: ANOVA/appropriate nonparametrics for group comparisons; repeated-measures ANOVA; Kaplan–Meier for flap survival; Pearson/Spearman for correlations. Two-sided alpha 0.05.

## 2. BACKGROUND AND RATIONALE

DIEP flap reconstruction avoids implants and offers natural contour, but intraoperative microcirculatory instability and I/R significantly affect outcomes, with reported double-digit rates of fat necrosis or partial flap loss. I/R triggers a burst of ROS (mitochondrial and enzyme sources such as xanthine oxidase and NOX), causing lipid peroxidation, apoptosis, endothelial dysfunction, and inflammation. Conventional ICG-NIR imaging assists real-time perfusion assessment, yet is constrained by limited depth and autofluorescence. NIR-IIb improves penetration and SNR, better capturing subcutaneous fat and deep microvasculature. Mn/QD-SAC integrates imaging with therapy: single-atom Mn active sites provide ROS-scavenging enzyme-mimetic activity while QDs enable NIR-IIb emission. Pilot evidence in a murine brain injury model supports feasibility for ROS suppression, inflammation inhibition, and tissue repair, warranting systematic evaluation in flap I/R models.

### 3. OBJECTIVES Primary

- (1) Develop and validate in vivo NIR-IIb imaging performance (sensitivity, timing, quantification) of Mn/QD-SAC in DIEP flap I/R and compare to ICG-NIR, laser Doppler/speckle, and tissue oxygenation measurements.
- (2) Demonstrate antioxidant, anti-inflammatory, and anti-apoptotic effects and mechanisms (e.g., Nrf2/HO-1, NF-κB, JAK/STAT).
- (3) Establish a feasible workflow in murine flap I/R and a clinical preclinical human biospecimen sub-study (DIEP patient peripheral blood) to inform future trials and safety assessment.

#### 4. STUDY DESIGN OVERVIEW

- (1) Part A: Materials synthesis and characterization of Mn/QD-SAC (physicochemical, optical, catalytic).
  - (2) Part B: In vitro mechanistic assays in endothelial, adipose/mesenchymal, and

immune cells under hypoxia-reoxygenation (H/R).

- (3) Part C: In vivo murine DIEP-like flap I/R model to test NIR-IIb imaging performance and therapeutic efficacy; safety and biodistribution.
- (4) Part D: Human biospecimen sub-study (observational) in DIEP patients for peripheral blood biomarkers at predefined perioperative timepoints; no investigational product administered to humans in this protocol.

#### 5. METHODS

- 5.1 Materials Synthesis and Characterization
- (1) Objective: Produce reproducible, stable Mn/QD-SAC and complete physicochemical, optical, and functional characterization.
- (2) QD preparation: Ag2Te/Ag2Se-based QDs with controlled size for NIR-IIb emission (1500–1700 nm).
- (3) Mn single-atom incorporation: Wet-chemical loading/thermal treatment to achieve isolated Mn sites on QD surfaces; confirm by HAADF-STEM.
- (4) Surface modification: mPEG-SH or DSPE-PEG ligand exchange/encapsulation to reduce protein adsorption and enhance circulation; measure zeta potential and solubility.
- (5) Characterization: TEM/HAADF-STEM, XPS, XRD, UV-Vis-NIR, and fluorescence spectroscopy (QY, emission peak), ESR for radical scavenging, and stability in serum/salt/protease.
- (6) In vitro catalytic activity: SOD-like and CAT-like assays; ESR trapping for •OH and O2•—.

## 5.2 In Vitro Models and Readouts

(1) Cell types:

Endothelial: HUVEC or HDMEC (barrier function, NO production, apoptosis).

Adipose/mesenchymal: hADSC; adipogenic 3T3-L1 (fat tissue susceptibility to I/R).

Immune: RAW264.7 (M1/M2 polarization, cytokine secretion).

- (2) H/R model: 1% O2 hypoxia for 4–8 h followed by reoxygenation (21% O2); monitor ROS dynamics and viability.
- (3) Groups: Vehicle; QD without Mn; Mn/QD-SAC low/medium/high doses; positive control NAC (e.g., 5 mM).
- (4) Readouts: Cell viability (CCK-8 or CellTiter-Glo), apoptosis (Annexin V/PI), ROS (DCFH-DA, MitoSOX), mitochondrial membrane potential (JC-1), cytokines (ELISA: TNF-α, IL-6, IL-1β), and Western blot (Nrf2, HO-1, p-NF-κB, p-STAT3, iNOS/Arg1).

# 5.3 In Vivo DIEP-like Flap I/R Model

- (1) Model: Murine abdominal perforator-based pedicled or free flap; define ischemia onset; two ischemia durations (2 h and 4 h) for mild/moderate injury.
- (2) Randomization (n≈8/group): Sham; I/R+PBS; I/R+QD (no Mn); I/R+Mn/QD-SAC low; I/R+Mn/QD-SAC medium; I/R+NAC.
- (3) Dosing (IV tail vein): Imaging 1 mg/kg; therapeutic 5 mg/kg; high-dose 10 mg/kg for toxicity arm.
  - (4) Timing: Administer at reperfusion; optional repeat at 6 h and 24 h.
- (5) Imaging: NIR-IIb intraoperative and at 0 min, 1 h, 6 h, 24 h, 72 h, Day 7, Day 14; record ROI intensity, perfused area, time-to-peak, SNR. Cross-validate with ICG-NIR

(intraop) and laser Doppler/speckle.

(6) Endpoints:

Functional/imaging: Flap survival area (Day 7-14), predictive accuracy of imaging vs

final survival.

Molecular/tissue: ROS and oxidative stress (MDA, 8-OHdG, 4-HNE), GSH/GSSG;

cytokines (tissue/serum ELISA); IHC (CD31, MPO, MMP-9); TUNEL; Western blot

(Nrf2, HO-1, p–NF-κB, p-STAT3).

Safety/biodistribution: CBC; serum chemistries (ALT/AST, creatinine); histopathology

(liver/kidney/spleen/lung/heart); ICP-MS of Ag and Mn in blood/organs.

(7) Blinding: Randomization of animals; imaging and histology analyses performed

blinded to group.

5.4 Human Biospecimen Sub-study (Observational)

(1) Population: Female, 18–70, undergoing immediate DIEP flap reconstruction after

breast cancer surgery; n≈30 convenience sample.

(2) Consent/IRB: Written informed consent before any procedures. Protocol and ICF

approved by the hospital ethics committee; amendments submitted for approval.

(3) Data and samples:

De-identified clinical data: age, BMI, operative time, ischemia duration, clinical flap

viability, complications.

Peripheral blood draws (10 mL each; serum tube + EDTA) at: pre-op baseline;

postoperative 0 h (immediate), 6 h, 24 h, and 72 h.

Analytes:

Hematology/coagulation: CBC, PT, APTT, fibrinogen, D-dimer.

Inflammation/oxidative stress: IL-6, IL-1β, TNF-α, IL-8/IL-10/IL-18, MDA, 8-iso-PGF2α, SOD, CAT, GSH-Px, total antioxidant capacity.

Injury/repair: Lactate, LDH, HMGB1, CK-MB, vWF, VEGF, HIF-1α.

Notes: Results are for research only and not used for clinical decision-making unless an incidental clinically actionable finding is identified and IRB-approved for disclosure.

#### 6. OUTCOME MEASURES

# Primary

- (1) In vivo therapeutic efficacy: Flap survival rate (%) at Day 7.
- (2) In vivo imaging: NIR-IIb SNR and correlation with final flap survival area.

# Secondary

- (1) Materials: Quantum yield; ROS scavenging efficiency; SOD-like and CAT-like activities.
  - (2) In vitro: Cell viability; apoptosis; ROS levels; cytokines; pathway proteins.
- (3) In vivo biology: MDA, SOD, GSH-Px; cytokines (TNF-α, IL-6, IL-1β, IL-10); histology scores; TUNEL; WB/IHC markers.
- (4) Safety: Body weight; CBC; chemistries; organ histopathology; elemental distribution/clearance (ICP-MS).

## 7. STATISTICAL ANALYSIS PLAN

- (1) Analysis populations: All randomized animals analyzed per assigned group. All processed biospecimens are included if predefined QC passes.
- (2) Descriptive statistics: Mean±SD or median[IQR] as appropriate; 95% CIs where informative.

- (3) Group comparisons: One-way ANOVA with post hoc tests (e.g., LSD-t) for parametric data; Kruskal–Wallis with Dunn's post hoc for nonparametric data.
- (4) Repeated measures: Repeated-measures ANOVA with appropriate covariance structure; Greenhouse–Geisser correction if sphericity is violated.
- (5) Survival analyses: Kaplan-Meier for flap survival; log-rank test for group differences.
  - (6) Correlations: Pearson (parametric) or Spearman (nonparametric).
  - (7) Multiplicity: Control via planned comparisons; exploratory nature acknowledged.
- (8) Sample size: Preclinical exploratory study; no formal power calculation. Group size  $n\approx8$  informed by prior effect sizes and feasibility. Human sub-study ( $n\approx30$ ) is hypothesis-generating.
  - (9) Software: SPSS v26.0 and GraphPad Prism v9.0.
  - (10) Significance: Two-sided alpha 0.05.

# 8. DATA MANAGEMENT AND QUALITY ASSURANCE

- (1) Data capture: De-identified unique study IDs. Source data is maintained securely.

  Double data entry or programmatic QC where feasible.
- (2) Monitoring: Periodic internal review of consent documentation, sample logs, imaging raw files, and analysis scripts.
- (3) Archiving: Retain per regulations; controlled destruction or extended retention with IRB approval.

### 9. PROTECTION OF HUMAN SUBJECTS AND PRIVACY

- (1) Consent and ethics: Clear explanation of purpose, procedures, risks/benefits; voluntary participation; IRB approval before initiation; amendments submitted for review.
- (2) Privacy: Coded IDs at collection; linkage file stored separately with restricted access. Publications use aggregate or anonymized data only.
- (3) Data security: Encrypted institutional servers; role-based access; regular backups; no public cloud for raw PHI. Paper records are stored locked.
- (4) Biospecimens: Labeled by ID only; used solely for prespecified assays. Residual samples require new IRB approval and/or renewed consent, or are destroyed per biosafety procedures.
- (5) Feedback: Individual lab results are not returned for clinical use unless incidental, clinically actionable findings are confirmed and IRB-approved for disclosure.

### 10. RISK-BENEFIT ASSESSMENT

- (1) Animals: Risks from surgery/anesthesia/agents mitigated by veterinary oversight and humane endpoints; analgesia per IACUC.
- (2) Human sub-study: Minimal risk from phlebotomy; no investigational product administered to humans in this protocol. Potential societal benefit from improved understanding of I/R biomarkers and imaging strategies.

### 11.ETHICAL AND REGULATORY COMPLIANCE

- (1) Conduct per Declaration of Helsinki, International Ethical Guidelines, and applicable national regulations and institutional policies.
  - (2) Animal studies per institutional IACUC standards and relevant guidelines.

#### 12.DISSEMINATION AND DATA SHARING

(1) Results will be disseminated in peer-reviewed publications and conferences.

(2) IPD sharing plan: No sharing of IPD is planned due to patient privacy and ethical

considerations, lack of consent for third-party data sharing, institutional/regulatory

restrictions, and limited resources for secure de-identification/hosting. Aggregate

results will be available in publications or upon request.

13. Administrative Information

Version: v1.0

Version Date: 11 Sep 2025.

Department: Breast Surgery, Hubei Cancer Hospital

Sponsor/Institution: Hubei Cancer Hospital